CLINICAL TRIAL: NCT03417323
Title: Effects of Compression Wear on Whole-body Electromyostimulation and Exercise-induced Muscle Soreness. A Randomized Controlled Trial.
Brief Title: Effects of Compression Wear on Muscle Soreness
Acronym: COMDOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Compression_DOMS_EMS
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Muscular Regeneration; Repeated Bout Effect of WB-EMS

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive garment (Experimental): Groups wear compression garment after WB-EMS induced muscle soreness
  Interventions: Other: Compression
- No compression garment (No Intervention): Groups wear no compression garment after WB-EMS induced muscle soreness

INTERVENTIONS:
Other: Compression — Participants in the treatment group wear compression garment after intense WB-EMS application for 24 h, and 12 h for day 2, 3, 4 post WB-EMS.
  Arms: Compressive garment

SUMMARY:
The study address two main topics:

1. The effect of compression garment on whole-body electromyostimulation (WB-EMS) induced muscle soreness in young adults
2. The repeated bout effect of one intense session of WB-EMS as determined by various regeneration parameters

DETAILED DESCRIPTION:
Using a cross-over design we applied 2 intense WB-EMS training sessions either with or without subsequent wearing of compression garments (long tights) for 5 days at baseline and after a washout period of 4 weeks. Healthy young to middle aged athletes used compression garments immediately postexercise for 24 hours and further 12 h during the day. Blood samples, questionnaires, resting metabolic rate and performance test were applied prior and 24, 48,72 and 96 h post-exercise consistently without wearing compression garments.

ELIGIBILITY:
Inclusion Criteria:

* healthy athletes with >5 years of experience in competition balls sports and corresponding discipline specific resistance exercise

Exclusion Criteria:

* diseases and medication affecting muscle metabolism
* contraindication for WB-EMS

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum isokinetic leg extensor strength | 5 days
  Changes of isokinetic leg extensor strength during the intervention period

SECONDARY OUTCOMES:
Perceived physical state | 5 days
  Changes of perceived physical state as determined by the WKV-scale (Kleinert, 2001) during the intervention period
Resting metabolic rate | 5 days
  Changes of resting metabolic rate during the intervention period
Myoglobin | 5 days
  Changes of myoglobin-levels during the intervention period
Heart rate variability | 5 days
  Changes of Heart rate variability during the intervention period
creatine-kinase (CK) concentration | 5 days
  Changes of CK-levels during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Lötzerich, PhD, Study Chair — German Sport University, Cologne; Wolfgang Kemmler, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School
Locations (2):
- Germany (2):
  - Institute of Medical Physics University of Erlangen-Nurnberg, Erlangen
  - Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kemmler W, Teschler M, Bebenek M, von Stengel S. [(Very) high Creatinkinase concentration after exertional whole-body electromyostimulation application: health risks and longitudinal adaptations]. Wien Med Wochenschr. 2015 Nov;165(21-22):427-35. doi: 10.1007/s10354-015-0394-1. Epub 2015 Oct 26. German. PMID 26498468
- See also: Institution homepage — http://www.imp.uni-erlangen.de/